CLINICAL TRIAL: NCT03397901
Title: Transverse Colostomy for Refractory Hemorrhagic Chronic Radiation Proctitis With Moderate to Severe Anemia: a Prospective Cohort Study
Brief Title: Transverse Colostomy for Refractory Hemorrhagic Chronic Radiation Proctitis: a Prospective Cohort Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lei Wang, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Colostomy-001
Record Dates: First submitted 2017-12-26; First posted 2018-01-12 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Chronic Radiation Proctitis; Rectal Bleeding; Colostomy Stoma; Anemia
Keywords: chronic radiation proctitis; rectal bleeding; transverse colostomy; refractory; moderate to severe anemia
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transverse colostomy (Experimental): Diverting transverse colostomy were conducted under general or epidural anesthesia in the operating room. The transverse colon was pulled out through one 2*2cm incision. The omentum was dissected from transverse colon, and a double-cavity stoma of transverse colon was then created.
  Interventions: Procedure: Transverse colostomy

INTERVENTIONS:
Procedure: Transverse colostomy — Transverse double-cavity colostomy

SUMMARY:
Refractory rectal bleeding of chronic radiation proctitis (CRP) is still problematic and does not respond to medical treatments including reagents, endoscopic argon plasma coagulation (APC) or topical formalin. We proposed this prospective cohort study, to assess the efficacy and safety of colostomy in treating refractory hemorrhagic CRP with moderate to severe anemia, to provide higher-quality evidence of colostomy in these patients.

DETAILED DESCRIPTION:
Chronic radiation proctitis (CRP) is a common complication after radiotherapy of pelvic malignancies, accounting for 5%-20% of cases. Rectal bleeding is the most common symptom, which accounts for > 80% of CRP patients. Mild to moderate bleeding can be controlled by medical agents like sucralfate, endoscopic argon plasma coagulation (APC) or topical formalin. Severe and refractory bleeding is still problematic and refractory to these above medical treatments. Our previous retrospective study found that colostomy obtained a higher rate of bleeding remission (94% vs 12%) in 6 months, especially in control of transfusion-dependent bleeding (100% vs0%), when compared to conservative treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed with pelvic malignancies, including gynecologic, prostate, or urinary cancers;
* History of pelvic radiation;
* No tumor recurrence or metastasis;
* Refractory hemorrhagic CRP;
* Time of rectal bleeding >6 months;
* SOBS=3 points;
* severe anemia （Hb≤7 g/dl）or transfusion history for CRP bleedings.

Exclusion Criteria:

* Severe complications of CRP, including deep ulcer or fistula, stricture, necrosis, refractory perianal pain;
* Other hemorrhagic diseases, like III-IV degree hemorrhoids;
* History of colon or rectum resection;
* Intestinal obstruction and surgery needed;
* with contraindications to general anaesthesia (ASA class 4 or 5);
* pregnant or breast-feeding;
* history of mental disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
remission rate of rectal bleeding after colostomy | 6 mon after colostomy
  retcal bleeding is assessed by soma scores

SECONDARY OUTCOMES:
Remission rate of rectal bleeding | 1 year, 2years, 3 years
  retcal bleeding is assessed by soma scores
Rate of colostomy closure | 1 years, 1.5 years, 2 years
  assess endoscopic findings before closure
Rate of severe CRP complications | 3 years
  include transfusion, deep ulceration or fistula, stricture, and refractory perianal pain
endoscopic score | 1 year
  Score of Vienna Rectoscopy Score (VRS)
endoscopic score | baseline, 6 months, 1 year, 2 years, 3 years
  Score of Rectal Telangiectasia Density
Quality of life by EORTC scores | baseline, 6 months, 1 year, 2 years, 3 years
  The European Organization for Research and Treatment of Cancer QLQ-C30 (EORTC QLQ-C30),The EORTC QLQ-C30 is a 30-item questionnaire composed of multi-item scales and single items that reflect the multidimensionality of the quality-of-life construct. It incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), and a global health and quality-of-life scale.
Anorectal function outcomes | baseline, 6 months, 1 year, 2 years, 3 years
  by Wexner score including 5 items: incontinence of solid stool, watery stool, gas, necessary of nursing pads, change of living habit
Rate of colostomy complications | baseline, 6 months, 1 year, 2 years, 3 years
  such as prolapse, edema, necrosis, retraction.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, Professor, Principal Investigator — Sixth Affiliated Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No
IPD is private information

REFERENCES:
- [Background] Yuan ZX, Ma TH, Wang HM, Zhong QH, Yu XH, Qin QY, Wang JP, Wang L. Colostomy is a simple and effective procedure for severe chronic radiation proctitis. World J Gastroenterol. 2016 Jun 28;22(24):5598-608. doi: 10.3748/wjg.v22.i24.5598. PMID 27350738
- [Background] Ma TH, Yuan ZX, Zhong QH, Wang HM, Qin QY, Chen XX, Wang JP, Wang L. Formalin irrigation for hemorrhagic chronic radiation proctitis. World J Gastroenterol. 2015 Mar 28;21(12):3593-8. doi: 10.3748/wjg.v21.i12.3593. PMID 25834325